CLINICAL TRIAL: NCT01453803
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intravenously and Intranasally in Patients With Parkinson's Disease
Brief Title: Study to Assess the Safety and Effects of Autologous Adipose-Derived SVF Cells in Patients With Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-PK-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Parkinson's Disease
Keywords: Liposuction; ADSC; ASC; stem cell; Parkinson's Disease; Parkinson's; therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Injection and Intanasal infusion of AD-SVF (Experimental): AD-SVF
  Interventions: Procedure: Harvesting and Implantation of Adipose-Derived Stem Cells

INTERVENTIONS:
Procedure: Harvesting and Implantation of Adipose-Derived Stem Cells — The adipose tissue specimen will be collected from the patient's abdomen or applicable region using a liposuction cannula. The adipose tissue is transferred to the laboratory for separation of the adipose tissue-derived stem cells, which are then transferred for catheter injection.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with Parkinson's Disease and clinical outcomes.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of Adipose-Derived Stromal Cells (ASC) implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered via catheter into the Vertebral Artery and intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Patient with current diagnosis of PD with motor complications (as confirmed by neurologist) as per the standard criteria and guidelines.
* Responsiveness to Levodopa or dopa agonist. This is defined as improvement between Off and On UPDRS by at least 33% of the Motor UPDRS.
* PD of Stage 2.5, 3 & 4 of HOEHN & YAHR staging.
* Stable Parkinsonian medications for the 60 days prior to the surgical therapy.
* MRI not showing gross atrophy or any other pathology of brain.
* Patients with score less than 19 for the Montgomery-Asberg Rating Scale (MADRS) for Depression.
* NO Significant cognitive impairment.MMSE > 21.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* History of intracranial surgeries or implantation of a device for Parkinson's disease two years prior to treatment.
* History of psychiatric disorders like schizophrenia or psychotic disorders.
* History of other malignancy, with the exception of treated cutaneous squamous cell or basal cell carcinoma, within 5 years.
* Contraindication for MRI
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis will be evaluated by an expert as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgement, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection being treated by antibiotics within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last two years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
UPDRS (UNIFIED PARKINSON'S DISEASE RATING SCALE)-Behavior | 3 months
  Improvement in Mentation, Behavior and mood in on and off position
Number of participants with adverse events | 1 week
UPDRS- Improvement in Activities of Daily Living | 3 months
UPDRS- Improvement in motor Examination | 3 months
  Values compared to baseline
UPDRS- MODIFIED HOEHN AND YAHR STAGING | 3 months
  Compared to baseline
UPDRS- SCHWAB AND ENGLAND ACTIVITIES OF DAILY LIVING SCALE | 3 months
UPDRS (UNIFIED PARKINSON'S DISEASE RATING SCALE)Behavior | 6 months
  Improvement in Mentation, Behavior and mood in on and off position
Number of participants with adverse events | 2 weeks
Number of participants with adverse events | 4 weeks
UPDRS- Improvement in Activities of Daily Living | 6 months
UPDRS- Improvement in motor Examination | 6 months
UPDRS- MODIFIED HOEHN AND YAHR STAGING | 6 months
UPDRS- SCHWAB AND ENGLAND ACTIVITIES OF DAILY LIVING SCALE | 6 months

SECONDARY OUTCOMES:
Reduction of Parkinson's medications | 3 months
Improvement in subjective symptoms: facial expression, gait, and freezing | 3 months
Reduction of Parkinson's medications | 6 months
Improvement in subjective symptoms: facial expression, gait, and freezing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided